CLINICAL TRIAL: NCT05546268
Title: A Phase 1/2 Study of Oral MRT-2359 in Patients With MYC-Driven and Other Selected Solid Tumors Including Lung Cancer and Diffuse B-Cell Lymphoma
Brief Title: Study of Oral MRT-2359 in Selected Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Monte Rosa Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRT-2359-001
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: NSCLC; SCLC; High Grade Neuroendocrine Cancer; DLBCL; L-MYC and N-MYC Amplified Solid Tumors; NSCLC With High or Low L-MYC or N-MYC Expression; HR-positive, HER2-negative Breast Cancer; Prostate Cancer
Keywords: Small Cell Lung Cancer; Non-Small Cell Lung Cancer; L-MYC Amplification; N-MYC Amplification; L-MYC expression; N-MYC expression; High-grade neuroendocrine; Diffuse Large B-Cell Lymphoma; Molecular glue degrader; Anti-tumor; GSPT1; HR-positive; HER2-negative; Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Lymphoma, Large B-Cell, Diffuse; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1 Dose Escalation (Experimental): Patients with NSCLC, SCLC, high-grade neuroendocrine cancer of any primary site, any solid tumors with L-MYC or N-MYC amplification, or DLBCL
  Interventions: Drug: Oral MRT-2359
- Phase 2 Expansion - NSCLC (Experimental): Patients with NSCLC with high or low L-MYC or N-MYC expression
  Interventions: Drug: Oral MRT-2359
- Phase 2 Expansion - SCLC (Experimental): Patients with SCLC
  Interventions: Drug: Oral MRT-2359
- Phase 2 Expansion - L-MYC or N-MYC amplified solid tumors (Experimental): Patients with L-MYC or N-MYC amplified solid tumors
  Interventions: Drug: Oral MRT-2359
- Phase 2 Expansion - HR-positive, HER2-negative breast cancer (Experimental): Patients with HR-positive, HER2-negative breast cancer in combination with fulvestrant
  Interventions: Drug: Oral MRT-2359
- Phase 2 Expansion - Prostate Cancer (Experimental): Patients with prostate cancer in combination with enzalutamide
  Interventions: Drug: Oral MRT-2359

INTERVENTIONS:
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359.
  Arms: Phase 1 Dose Escalation
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359.
  Arms: Phase 2 Expansion - NSCLC
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359.
  Arms: Phase 2 Expansion - SCLC
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359.
  Arms: Phase 2 Expansion - L-MYC or N-MYC amplified solid tumors
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359 in conjunction with intramuscular administration of fulvestrant.
  Arms: Phase 2 Expansion - HR-positive, HER2-negative breast cancer
Drug: Oral MRT-2359 — Orally administered tablets of MRT-2359 in conjunction with orally administered enzalutamide.
  Arms: Phase 2 Expansion - Prostate Cancer

SUMMARY:
This Phase 1/2, open-label, multicenter study is conducted in patients with previously treated selected solid tumors, including non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), high-grade neuroendocrine cancer of any primary site, diffuse large B-cell lymphoma (DLBCL), and tumors with L-MYC or N-MYC amplification. Patients receive escalating doses of a GSPT1 molecular glue degrader MRT-2359 to determine safety, tolerability, maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of MRT-2359. Once the MTD and/or RP2D is identified, additional patients enroll to Phase 2 study, which includes molecular biomarkers stratification or selection, namely expression or amplification of L-MYC and N-MYC genes, hormone receptor positive (HR)-positive, human epidermal growth factor 2 (HER2)-negative breast cancer and prostate cancer.

DETAILED DESCRIPTION:
This Phase 1/2, open-label, multicenter, dose escalation and expansion study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and preliminary clinical activity of MRT-2359 in patients with previously treated selected solid tumors, including lung cancer (NSCLC and SCLC), high-grade neuroendocrine cancer of any primary site, and DLBCL.

* The primary aim of Phase 1 part is safety, tolerability, MTD and/or RP2D of MRT-2359.
* The primary aim of Phase 2 part is assessment of preliminary anti-tumor activity of MRT-2359.

ELIGIBILITY:
Phase 1 enrollment population:

* NSCLC
* SCLC
* High-grade neuroendocrine cancer of any primary site
* Any solid tumors with L-MYC or N-MYC amplification
* DLBCL

Phase 2 enrollment population:

* Any solid tumors with L-MYC or N-MYC amplification
* NSCLC with high or low L-MYC or N-MYC expression status (testing will be provided) or SCLC
* HR-positive, HER2-negative breast cancer - MRT-2359 in combination with fulvestrant
* Non-neuroendocrine prostate cancer - MRT-2359 in combination with enzalutamide

Phase 1 and Phase 2 Inclusion Criteria:

* Have a selected advanced solid tumor or DLBCL (listed above) for which there are no further standard therapeutic options available
* Be age ≥ 18 years and willing to voluntarily complete the informed consent process
* A predicted life expectancy of ≥ 3 months and an ECOG performance status ≤ 2
* Have measurable disease by RECIST 1.1 (Eisenhauer et al., 2009) in case of solid tumors or Revised Response Criteria for Malignant Lymphoma (Phase 1 only) (Cheson et al., 2014) in case of DLBCL
* Have adequate organ function defined by the selected laboratory parameters
* If female of childbearing potential, avoid becoming pregnant and agree to use acceptable methods of contraception after informed consent, throughout the study, and for 90 days after the last dose of MRT-2359
* Male of reproductive potential must use an approved methods of contraception from informed consent until 90 days after study discharge

Exclusion Criteria:

* Have received prior chemotherapy, definitive radiation, biological cancer therapy or any investigational agent within 21 days before the first dose of study treatment, or have any AEs that have failed to recover to baseline. In patients with prostate cancer, continuance of systemic therapies to maintain castration levels of testosterone is allowed. Pre-menopausal patients with hormone-dependent breast cancer can continue on therapies used for suppression of ovarian function.
* Have received bisphosphonates or denosumab within 14 days before the first administration of the study drug unless they were given for acute hypercalcemia
* Inability to swallow oral medication
* Have received prior therapy with a GSPT1 degrader that was discontinued due to an AE
* Have received prior auto-HCT and not fully recovered from effects of the last transplant
* Have received prior allogeneic hematopoietic stem cell transplantation within past 6 months and/or have symptoms of graft-versus-host disease. Patients requiring minimal intervention such as topical steroids are eligible
* Have received a live vaccine within 90 days before the first dose of study treatment
* COVID-19 immunization within 14 days of receiving the first dose of MRT-2359
* Current use of chronic systemic steroid therapy in excess of replacement doses (prednisone ≤ 10 mg/day is acceptable)
* Have clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug
* Have a history of a second malignancy, unless controlled not requiring therapy
* Have clinically active central nervous system involvement and/or carcinomatous meningitis. Patients with treated and stable brain metastases (not progressing for at least 4 weeks prior to enrollment) not requiring steroids are eligible
* Have a confirmed history of (non-infectious) pneumonitis that required steroids
* Have known human immunodeficiency virus (HIV) unless the patient is on antiviral therapy with undetectable HIV RNA levels
* Have known hepatitis B or C infection(s) unless treated with undetectable hepatitis B DNA or hepatitis C RNA levels
* Clinically significant cardiac disease
* Be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Evaluates safety and tolerability of MRT-2359 over a 28-day cycle by the occurrence and frequency of dose limiting toxicities (DLTs) for determination of the MTD and/or RP2D | 28 days
Phase 2 Evaluates preliminary anti-tumor activity of MRT-2359 by overall response rate (ORR) as determined by RECIST 1.1 | 56 days (up to approximately 24 months from screening to end of study participation

SECONDARY OUTCOMES:
Phase 1 safety and tolerability of MRT-2359 (orally over a 28-day cycle) by the nature, incidence, and severity of all treatment-emergent adverse events (TEAEs), including treatment-related TEAEs and serious adverse events (SAEs) | 18 months
Phase 1 preliminary anti-tumor activity: ORR (RECIST 1.1/Revised Response Criteria for Malignant Lymphoma),duration of response for complete response(CR)/partial response(PR), disease control rate, progression-free survival, overall survival | 18 months
Phase 1 Dose Escalation characterizes the PK profile of MRT-2359 by standard primary PK parameters including, but not limited to, AUC, Cmax, tmax, and t1/2 | 28 days
Phase 1 Dose Escalation evaluates the effect of a high-fat meal on the relative bioavailability of MRT-2359 by standard primary PK parameters including, but not limited to, AUC and Cmax | 7 days
Phase 2 Dose Expansion evaluates the safety and tolerability of MRT-2359 administered orally over a 28-day cycle by the nature, incidence, and severity of all TEAEs, including treatment-related TEAEs and SAEs according to the NCI CTCAE, version 5.0 | 24 months
Phase 2 Dose Expansion evaluates additional measures of the preliminary anti-tumor activity of MRT-2359 such as DoR (in patients with the best overall response of CR or PR) | 24 months
Phase 2 Dose Expansion further characterizes the PK profile of MRT-2359 by evaluating MRT-2359 plasma concentration to establish PK parameters including, but not limited to, Cmax, tmax, AUC0-t, AUC0inf, mean residence time, accumulation ratio, etc. | 28 days
Phase 2 Dose Expansion evaluates additional measures of the preliminary anti-tumor activity of MRT-2359 such as DCR | 24 months
Phase 2 Dose Expansion evaluates additional measures of the preliminary anti-tumor activity of MRT-2359 such as PFS | 24 months
Phase 2 Dose Expansion evaluates additional measures of the preliminary anti-tumor activity of MRT-2359 such as OS | 24 months
Phase 2 Dose Expansion evaluates additional measures of the preliminary anti-tumor activity of MRT-2359 such as PSA response | 24 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Sarah Cannon Research Institute, Lake Mary, Florida
  - Indiana University, Bloomington, Indiana
  - University of Kansas Cancer Center, Lawrence, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Irving Medical Centre, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START) Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists Research Institute, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No